CLINICAL TRIAL: NCT00012974
Title: Innovative Strategies for Implementing New CHF Guideline Recommendations
Brief Title: Telephone Administered Psychotherapy for the Treatment of Depression for Veterans in Rural Areas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHI 99-063
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Heart Failure; Beta-blocker Treatment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: GTelephone-administered Cognitive-Behavioral Therapy (T-CBT); Procedure: Provider education, computer reminders, nurse case management

INTERVENTIONS:
Behavioral: GTelephone-administered Cognitive-Behavioral Therapy (T-CBT)
Procedure: Provider education, computer reminders, nurse case management

SUMMARY:
The purpose of this study is to examine the efficacy of telephone-administered cognitive-behavioral therapy (T-CBT) in treating major depression among veterans served by community-based outpatient clinics (CBOCs) in the Veteran�s Integrated Service Network (VISN) 21, which serves rural areas in Northern California

DETAILED DESCRIPTION:
More that 20% of patients in primary care have depressive disorders. While primary care is the principal venue for treatment for depression, fewer than 25% of depressed patients receive adequate treatment for their depression. These outcomes can be worse when there are barriers to treatment such as living in a rural area. Several studies have found that given a choice, about two-thirds of depressed primary care patients prefer psychotherapy or counseling over antidepressant medication.

This is a controlled, randomized trial in which subjects meeting criteria for major depressive disorder (MDD) from primary care settings in VISN 21 including CBOCs will be randomly assigned to one of two conditions: 1) a 16-session manualized telephone administered cognitive behavioral therapy (T-CBT) delivered over 24 weeks or 2) a treatment-as-usual (TAU) condition. Telephone-administered cognitive behavioral therapy (T-CBT) is an intervention aimed at improving coping skills and social functioning. It is divided into two phases: 1) an initial treatment phase consisting of 12 weekly sessions aimed at reducing symptoms of depression, and 2) a booster phase in which 4 sessions are provided at increasingly greater intervals to target maintenance of treatment gains. T-CBT, administered by doctoral level psychologists, will be compared to a treatment-as-usual (TAU) condition that controls for the natural course of depression during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must have chronic heart failure, systolic left ventricular dysfunction (ejection fraction less than or equal to 45%), not be receiving beta-blockers, and not have contraindications to beta-blockers.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Reduction in severity of depression; scores on depression rating scales at baseline, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Maintenance of treatment gains at 6 month follow-up (week 48).

CONTACTS AND LOCATIONS:
Overall Officials: Barry M Massie, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

REFERENCES:
- [Result] Massie BM. Comment--LVADs as long-term cardiac replacement: Success but on what terms and at what cost? J Card Fail. 2002 Apr;8(2):61-2. doi: 10.1054/jcaf.2002.33167. No abstract available. PMID 12016627
- [Result] Cuffe MS, Califf RM, Adams KF Jr, Benza R, Bourge R, Colucci WS, Massie BM, O'Connor CM, Pina I, Quigg R, Silver MA, Gheorghiade M; Outcomes of a Prospective Trial of Intravenous Milrinone for Exacerbations of Chronic Heart Failure (OPTIME-CHF) Investigators. Short-term intravenous milrinone for acute exacerbation of chronic heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1541-7. doi: 10.1001/jama.287.12.1541. PMID 11911756
- [Result] Leier CV, Silver MA, Massie BM, Young JB, Fowler MB, Ventura HO, Hershberger RE. Nuggets, pearls, and vignettes of master heart failure clinicians. Part 1--the medical history. Congest Heart Fail. 2001 Sep-Oct;7(5):245-249. doi: 10.1111/j.1527-5299.2001.00307.x. No abstract available. PMID 11832662
- [Result] Dauterman KW, Go AS, Rowell R, Gebretsadik T, Gettner S, Massie BM. Congestive heart failure with preserved systolic function in a statewide sample of community hospitals. J Card Fail. 2001 Sep;7(3):221-8. doi: 10.1054/jcaf.2001.26896. PMID 11561221
- [Result] Go AS, Rao RK, Dauterman KW, Massie BM. A systematic review of the effects of physician specialty on the treatment of coronary disease and heart failure in the United States. Am J Med. 2000 Feb 15;108(3):216-26. doi: 10.1016/s0002-9343(99)00430-1. PMID 10723976
- [Result] Cuffe MS, Califf RM, Adams KF, Bourge RC, Colucci W, Massie B, O'Connor CM, Pina I, Quigg R, Silver M, Robinson LA, Leimberger JD, Gheorghiade M. Rationale and design of the OPTIME CHF trial: outcomes of a prospective trial of intravenous milrinone for exacerbations of chronic heart failure. Am Heart J. 2000 Jan;139(1 Pt 1):15-22. doi: 10.1016/s0002-8703(00)90303-x. PMID 10618557
- [Result] Massie BM. Obesity and heart failure--risk factor or mechanism? N Engl J Med. 2002 Aug 1;347(5):358-9. doi: 10.1056/NEJMe020065. No abstract available. PMID 12151474
- [Result] Massie BM, Armstrong PW, Cleland JG, Horowitz JD, Packer M, Poole-Wilson PA, Ryden L. Toleration of high doses of angiotensin-converting enzyme inhibitors in patients with chronic heart failure: results from the ATLAS trial. The Assessment of Treatment with Lisinopril and Survival. Arch Intern Med. 2001 Jan 22;161(2):165-71. doi: 10.1001/archinte.161.2.165. PMID 11176729
- [Result] Ashton CM, Bozkurt B, Colucci WB, Kiefe CI, Mann DL, Massie BM, Slawsky MT, Tierney WM, West JA, Whellan DJ, Wray NP. Veterans Affairs Quality Enhancement Research Initiative in chronic heart failure. Med Care. 2000 Jun;38(6 Suppl 1):I26-37. doi: 10.1097/00005650-200006001-00004. PMID 10843268
- [Result] Gottlieb SS, Abraham W, Butler J, Forman DE, Loh E, Massie BM, O'connor CM, Rich MW, Stevenson LW, Young J, Krumholz HM. The prognostic importance of different definitions of worsening renal function in congestive heart failure. J Card Fail. 2002 Jun;8(3):136-41. doi: 10.1054/jcaf.2002.125289. PMID 12140805
- [Result] Massie BM. Treating heart failure: it's time for new paradigms and novel approaches. J Card Fail. 2002 Jun;8(3):117-9. doi: 10.1054/jcaf.2002.126485. No abstract available. PMID 12140801
- [Result] Ansari M, Tutar A, Bullard J, Teerlink J, Massie B. Cardiology specialist care of heart failure patients improves survival. [Abstract]. Journal of the American College of Cardiology. 2001 Jun 1; 37:189A.
- [Result] Massie BM. Neurohormonal blockade in chronic heart failure. How much is enough? Can there be too much? J Am Coll Cardiol. 2002 Jan 2;39(1):79-82. doi: 10.1016/s0735-1097(01)01715-6. No abstract available. PMID 11755290
- [Result] Ansari M, Tutar A, Bullard J, Teerlink J, Massie B. Heart failure in a veteran cohort: Predictors of outcome. [Abstract]. Journal of the American College of Cardiology. 2001 Jun 1; 37:1581.
- [Result] Frances CD, Noguchi H, Massie BM, Browner WS, McClellan M. Are we inhibited? Renal insufficiency should not preclude the use of ACE inhibitors for patients with myocardial infarction and depressed left ventricular function. Arch Intern Med. 2000 Sep 25;160(17):2645-50. doi: 10.1001/archinte.160.17.2645. PMID 10999979
- [Result] Massie BM. The year in heart failure: 2004. J Card Fail. 2005 Feb;11(1):1-6. doi: 10.1016/j.cardfail.2005.01.001. No abstract available. PMID 15704055
- [Result] Massie BM. Isosorbide dinitrate plus hydralazine was effective for advanced heart failure in black patients. ACP J Club. 2005 Mar-Apr;142(2):37. No abstract available. PMID 15739984
- [Result] Teerlink JR, Massie BM. Nesiritide and worsening of renal function: the emperor's new clothes? Circulation. 2005 Mar 29;111(12):1459-61. doi: 10.1161/01.CIR.0000160874.48045.54. No abstract available. PMID 15795361
- [Result] Massie BM. Heart failure trials: are they becoming impractical? J Card Fail. 2005 Apr;11(3):161-3. doi: 10.1016/j.cardfail.2005.03.001. No abstract available. PMID 15812741